CLINICAL TRIAL: NCT03852121
Title: Bibliotherapy for Improving Caregiving Appraisal Among Informal Caregivers of People With Dementia: A Pilot Randomized Controlled Trial
Brief Title: Bibliotherapy for Improving Caregiving Appraisal Among Informal Caregivers of People With Dementia: A Pilot RCT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr Daphne Cheung, Principal Investigator, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20181120001
Record Dates: First submitted 2019-02-04; First posted 2019-02-25 (Actual); Last update posted 2020-10-19 (Actual); Status verified 2020-10

CONDITIONS: Dementia
Keywords: caregiving appraisal; bibliotherapy; psychological wellbeing; informal caregiver
MeSH Terms: conditions — Dementia | interventions — Bibliotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Participants will receive bibliotherapy without withdrawing from the usual care. They will be asked to read the designated manual (consists of eight chapters) within a recommended period of time (over 8 weeks). Weekly telephone coaching will also be provided to figure out participants understanding, find out the unsolved problems and guide them for finding out the solution by themselves. An orientation will be organized before the first session. Two booster sessions will be organized during the study.
  Interventions: Behavioral: Bibliotherapy
- Control group (No Intervention): The participants in the control group will only receive usual care provided by the community health professionals.

INTERVENTIONS:
Behavioral: Bibliotherapy — Bibliotherapy is the use of reading materials for therapeutic benefits. In this study, an evidence-based modified manual will be used as the reading material. The manual adopts the self-directed problem-solving approach to dementia caregiving, examples of how other caregivers solve the specific problem for each chapter is included in the corresponding chapter. Bibliotherapy also involves guided learning by reading written information, enabling caregivers to solve their caregiving problems "step-by-step", so telephone coach is designed to figure out participants understanding, find out the unsolved problems and guide them for finding out the solution by themselves.
  Arms: Intervention group

SUMMARY:
This is a 8-week pilot randomized controlled trial utilizing bibliotherapy compared with usual care to investigate the feasibility and acceptability of bibliotherapy among informal caregivers of people with dementia in China, and preliminarily examine the efficacy on improving caregiving appraisal.

DETAILED DESCRIPTION:
Background: China is one of the countries with the highest number of people with dementia (PWD), while over 90% of PWD are cared by informal caregivers in the community. Informal caregivers are found to have higher level of stress, and lower level of well-being than non-caregivers. However, positive outcomes of caregiving have also been noted. Caregiving appraisal is caregivers' cognitive evaluation of potential caregiving stressors and the efficacy of their coping efforts related to caregiving experience. Based on Lawton's Caregiving Appraisal and Psychological Well-being Model, caregiving appraisal is an important factor that leads to the positive or negative well-being outcomes of caregivers. Addressing the caregiving appraisal of informal caregiver may be able to help in promoting the caregiver well-being and delay premature institutionalization. Intervention for improving dementia caregiving appraisal is still scarce, especially in China. Bibliotherapy is the process of learning from high-quality written materials for therapeutic benefits, it has been proved to be effective in improving caregiving appraisal of informal caregivers of people with psychosis and depression, its effect on dementia caregivers is unsure.

Objectives: There are two research objectives in this study: (1) To determine the feasibility and acceptability of the evidence-based bibliotherapy protocol among informal caregivers of PWD in China. (2) To preliminarily explore the efficacy of bibliotherapy on improving caregiving appraisal.

Methods:

Sixty participants will be recruited from Zhengzhou, China, and will be randomly allocated to either the intervention group or usual care group. The feasibility of the intervention will be explored in terms of the ease of participant recruitment, attendance rate and the attrition rate. The acceptability will be explored by interviews of participants in the intervention group at post-intervention. The Chinese version of Caregiving Appraisal Scale, the Chinese version of Ways of Coping Questionnaire, the Chinese version of Positive Aspects of Caregiving Scale, the Chinese version of Ryff's Psychological Well-being Scale, Alzheimer's Disease Knowledge Scale and Dementia Attitude Scale will be used to measure caregiving appraisal, coping, positive aspects of caregiving, psychological well-being, knowledge of dementia and attitude toward dementia of informal caregivers of PWD respectively. Descriptive statistics, Chi-square test, Mann Whitney U test, and independent t-test will be used to describe the participants' characteristics and compare the difference between groups at baseline. GEE will be used to examine the intervention efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Caregiver who provides regular care to a person with early to moderate level of any type of medical diagnosis of dementia (PWD) for at least 5 hours per week for at least 6 months;
* Aged 18 or above;
* Not paid for the care provided;
* Assist with at least one of PWD's daily activities;
* Be able to read;
* Can be contacted by phone.

Exclusion Criteria:

* Caregivers with unstable physical or mental conditions;
* Those with cognitive impairment;
* Those involved in another interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2020-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in caregiving appraisal | At baseline, immediate post intervention
  To be measured with the Chinese version of Caregiving Appraisal Scale (CAS). The Chinese version of CAS includes 26 items, divided into 4 subscales: caregiving burden, caregiving satisfaction, caregiving mastery, and caregiving impact. This is a 5 point Likert scale (1 = disagree a lot to 5 = agree a lot). The total score ranges from 26 to 130, with higher scores indicate more positive caregiving appraisal. The Cronbach's α for each subscale was 0.68~0.87.

SECONDARY OUTCOMES:
Changes in caregiver's coping | At baseline, immediate post intervention
  To be measured with the Chinese version of Ways of Coping Questionnaire. This questionnaire includes 20 items, divided into 2 subscales: the active coping subscale and the passive coping subscale. The passive coping subcale was recoded. The total score ranges from 0-60, higher score indicates more positive coping. It is a 4 point Likert scale (0 = never to 3 = often). The Cronbach's α was 0.90, αs for the two subscales were 0.89 and 0.78.
Changes in caregiver's psychological well-being | At baseline, immediate post intervention
  To be measured with the shorter Chinese version for Ryff's Psychological Well-being Scale. This scale includes 18 items, and is divided into 6 subscales: positive relations with others, autonomy, environmental mastery, personal growth, purpose in life and self-acceptance. This scale is a Likert 6 point scale, with 1 = strongly disagree to 6 = totally agree, higher scores indicate better psychological well-being. The total score ranges from 6-108. The scale has been tested in middle-aged and older people, the Cronbach's α was 0.92 for the total scale, and at least 0.60 for each subscale.
Changes in positive aspects of caregiving | At baseline, immediate post intervention
  To be measured with the Chinese version of Positive Aspects of Caregiving (C-PAC) Scale. It is a Likert 5 point scale ranging from 1 (strongly disagree) to 5 (strongly agree) regarding the extent to which providing care to their relatives with dementia had enabled them "feel important", "feel appreciated" etc. The scale has 11 items, divided into two subscales: enriching life and affirming self. The total score ranges from 5-55. The Cronbach's α was 0.89 for the total scale, the αs for enriching life and affirming self subscales were 0.85 and 0.84 respectively.
Changes in knowledge of dementia | At baseline, immediate post intervention
  To be measured with the Chinese version of Alzheimer's Disease Knowledge Scale. This scale has 30 items, with "true" or "false" choices for each item. The total score ranges from 0-30. Higher score indicates more knowledgement about dementia. The Cronbach's a was 0.785.
Changes in attitude toward dementia | At baseline, immediate post intervention
  To be measured with the Chinese version of Dementia Attitude Scale. This is a 20-item Likert 7 point scale (1=strongly disagree, 7=strongly agree). The total score ranges from 20-140, higher scores indicate more positive attitude toward dementia. The Cronbach's α was 0.818.

CONTACTS AND LOCATIONS:
Overall Officials: Daphne Cheung, PhD, Principal Investigator — School of Nursing, The Hong Kong Polytechnic University
Locations (1):
- School of Nursing, The Hong Kong Polytechnic University, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arain M, Campbell MJ, Cooper CL, Lancaster GA. What is a pilot or feasibility study? A review of current practice and editorial policy. BMC Med Res Methodol. 2010 Jul 16;10:67. doi: 10.1186/1471-2288-10-67. PMID 20637084
- [Background] Bilich LL, Deane FP, Phipps AB, Barisic M, Gould G. Effectiveness of bibliotherapy self-help for depression with varying levels of telephone helpline support. Clin Psychol Psychother. 2008 Mar-Apr;15(2):61-74. doi: 10.1002/cpp.562. PMID 19115429
- [Background] Campbell LF, Smith TP. Integrating self-help books into psychotherapy. J Clin Psychol. 2003 Feb;59(2):177-86. doi: 10.1002/jclp.10140. PMID 12552626
- [Background] Folkman, S., & Lazarus, R. S. (1988). Ways of coping questionnaire: Consulting Psychologists Press.
- [Background] Hsiao HY, Liu Z, Xu L, Huang Y, Chi I. Knowledge, Attitudes, and Clinical Practices for Patients With Dementia Among Mental Health Providers in China: City and Town Differences. Gerontol Geriatr Educ. 2016 Oct-Dec;37(4):342-358. doi: 10.1080/02701960.2014.990152. Epub 2015 Jan 27. PMID 25625718
- [Background] Lawton MP, Kleban MH, Moss M, Rovine M, Glicksman A. Measuring caregiving appraisal. J Gerontol. 1989 May;44(3):P61-71. doi: 10.1093/geronj/44.3.p61. PMID 2715587
- [Background] Lawton MP, Moss M, Kleban MH, Glicksman A, Rovine M. A two-factor model of caregiving appraisal and psychological well-being. J Gerontol. 1991 Jul;46(4):P181-9. doi: 10.1093/geronj/46.4.p181. PMID 2071844
- [Background] Lazarus, R. S., & Folkman, S. (1986). Stress, appraisal, and coping. New York: pringer.
- [Background] Li, R.-H. (2014). Reliability and validity of a shorter Chinese version for Ryff's psychological well-being scale. Health Education Journal, 73(4), 446-452.
- [Background] Lou VW, Lau BH, Cheung KS. Positive aspects of caregiving (PAC): scale validation among Chinese dementia caregivers (CG). Arch Gerontol Geriatr. 2015 Mar-Apr;60(2):299-306. doi: 10.1016/j.archger.2014.10.019. Epub 2014 Nov 7. PMID 25488014
- [Background] Sclan SG, Reisberg B. Functional assessment staging (FAST) in Alzheimer's disease: reliability, validity, and ordinality. Int Psychogeriatr. 1992;4 Suppl 1:55-69. doi: 10.1017/s1041610292001157. PMID 1504288
- [Background] Shechtman, Z. (2009). Bibliotherapy as a Method of Treatment. In Treating Child and Adolescent Aggression Through Bibliotherapy (pp. 1-17).
- [Background] Wang S, Cheung DSK, Leung AYM. Overview of dementia care under the three-tier long-term care system of China. Public Health Nurs. 2019 Mar;36(2):199-206. doi: 10.1111/phn.12573. Epub 2018 Dec 13. PMID 30549090
- [Background] Zheng X, Chung JO, Woo BK. Exploring the Impact of a Culturally Tailored Short Film in Modifying Dementia Stigma Among Chinese Americans: A Pilot Study. Acad Psychiatry. 2016 Apr;40(2):372-4. doi: 10.1007/s40596-015-0397-7. Epub 2015 Aug 26. PMID 26307362

DOCUMENTS (1):
  • Informed Consent Form (2018-12-01): https://cdn.clinicaltrials.gov/large-docs/21/NCT03852121/ICF_000.pdf